CLINICAL TRIAL: NCT06866015
Title: The Impact of an Activation-Socialisation Intervention Programme on the Emotionality and Loneliness of Older Adults in Slovak Elderly Care Facilities - a Pilot Study
Brief Title: Activation Programme's Impact on Seniors' Emotionality and Loneliness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diana Ďuricová (Other)
Responsible Party: Sponsor-Investigator, Diana Ďuricová, Principal Investigator, Matej Bel University
Organization: Matej Bel University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 162/2025
Record Dates: First submitted 2025-02-24; First posted 2025-03-10 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Emotional States; Loneliness; Seniors
Keywords: older adult; elderly care facilities; intervention programme; emotions; loneliness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Activation-socialization interventiom programme (Experimental)
  Interventions: Other: Activation-socialization intervention programme

INTERVENTIONS:
Other: Activation-socialization intervention programme — The proposed A-S IP (Author, 2021) includes 40 activities of three domains focusing mainly on the social-psychological level of education: the Laughter Therapy Concept (13), the Reminiscence Therapy Concept (13), and the Cognitive and Social Skills Stimulation Intervention Concept (14).
  The implementation of the A-S IP activities was designed for a time period of four weeks during weekdays. In the Hriňovčan care facility for older adults, mainly in the common room, two activities were implemented daily during the morning and afternoon hours reserved for this purpose. Morning activities (active) were from 10:00 to 11:00 a.m., and afternoon activities (passive) were from 1:00 to 2:00 p.m. The application of the activities was strictly determined and organised according to a time-thematic schedule that applied rules. The participants participated in group activities, and their participation was voluntary.

SUMMARY:
The goal of this pilot study is to verify the short-term effectiveness of the Activation-Socialisation Intervention Programme (A-S IP) on the psychosocial survival of older adults in a specific care facility. The main questions it aims to answer are:

* Does the A-S IP reduce the rate of negative emotional states in older adults?
* Does the A-S IP increase the rate of positive emotional states in older adults?
* Does the A-S IP reduce feelings of loneliness in older adults? Researchers will compare the experimental group (older adults participating in the A-S IP) to a control group (older adults not participating in the intervention) to assess the impact on emotional states and loneliness.

Participants will:

* Participate in 40 activities based on three domains (Laughter Therapy, Reminiscence Therapy, and Cognitive and Social Skills Stimulation)
* Engage in group activities for four weeks, with daily sessions scheduled in the morning and afternoon
* Provide feedback on their experiences through surveys and questionnaires to assess their emotional states and satisfaction with the intervention

The study will also explore whether the intervention contributes to the well-being of older adults, as measured by changes in their emotional states and feelings of loneliness.

DETAILED DESCRIPTION:
The study was registered retrospectively due to limited awareness of the registration requirement for behavioral interventions at the time of study initiation (in 2021). Initially, the research was designed as an exploratory study on a smaller scale, and the registration of a formal trial was not considered necessary.

As an early-career researcher and doctoral student, I was not initially aware of the necessity of registering behavioral intervention studies. However, as the study progressed and its significance became evident, I came to understand the importance of this process. Once I became aware of the registration requirements, I took the necessary steps to complete it accordingly.

Despite the late registration, the study was conducted according to a pre-specified protocol, with all methodological and ethical standards strictly adhered to (approved, for example, by the Ethics Committee of UMB). The hypotheses, study design, and analysis plan were defined prior to data collection, ensuring the integrity and transparency of the research.

ELIGIBILITY:
Inclusion Criteria:

* long-term residence in the facility,
* age over 62,
* willingness to participate,
* ability to participate (no severe cognitive or physical impairments)

Exclusion Criteria:

* significant physical problems,
* significant mental health problems,
* unwillingness to participate

Min Age: 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
the Scale of Emotional Habitual Subjective Well-being - SEHP (Džuka & Dalbert, 2002) | one month
  The Scale of Emotional Habituation of Subjective Well-Being - SEHP (Džuka & Dalbert, 2002) was used to examine the short-term effectiveness of the intervention programme. The self-esteem scale maps the frequency of experiencing positive and negative emotions, totalling 10. Negative emotional experiencing consists of six emotions such as anger, guilt, fear, pain, sadness, and shame, positive emotional experiencing consists of pleasure, physical freshness, joy, and happiness. The participants responded on a six-point scale (6 - almost always; 1 - almost never). The total score of negative emotions is the sum of negative emotions, and the total score of positive emotions is the sum of positive emotions (Džuka et al., 2021). An additional variable, loneliness, was added to the scale. It was assessed on an identical six-point scale.
  Unit of Measure: Score (Total score for positive and negative emotions)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Ďuricová, PhDr., Principal Investigator — Matej Bel University; Lenka Ďuricová, doc., Mgr., PhD., Study Director — Matej Bel University
Locations (1):
- Hriňovčan care facility for older adults, Hriňová, Slovakia, Slovakia

IPD SHARING:
Plan to Share IPD: No